CLINICAL TRIAL: NCT00753337
Title: The ACTIVE (Use of the Assurant® Cobalt Iliac Stent System in the Treatment of Iliac Vessel Disease) Study Using the Medtronic Assurant Cobalt Iliac Balloon-Expandable Stent System
Brief Title: The ACTIVE (Use of the Assurant® Cobalt Iliac Stent System in the Treatment of Iliac Vessel Disease) Study
Acronym: ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP085
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assurant Cobalt Iliac Stent (Experimental): Assurant® Cobalt Iliac Stent System
  Interventions: Device: Assurant® Cobalt Iliac Stent System

INTERVENTIONS:
Device: Assurant® Cobalt Iliac Stent System — Iliac Stenting

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the Assurant Cobalt Iliac Stent System in the treatment of de novo and restenotic lesions in iliac arteries of subjects with Peripheral Artery Disease (PAD).

DETAILED DESCRIPTION:
This study is being conducted to collect 9 month safety and efficacy data on the Assurant Cobalt Iliac Stent for all subjects enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* The lesion(s) is either de novo or restenotic in nature, located in the common iliac artery and/or the external iliac artery;
* The subject is symptomatic (Fontaine stage II or III) with a target lesion stenosis ≥ 50% .
* The target vessel(s) reference diameter is ≥ 6 mm and ≤ 10 mm by visual estimate;
* The lesion length is < 100 mm (10 cm)

Exclusion Criteria:

* Excessive peripheral vascular disease(PVD), unresolved fresh thrombus or tortuousity,or heavily calcified.
* Tissue loss in the target extremities.
* The target lesion is in a prosthetic vascular bypass graft or within 1 cm of a graft anastomosis;
* The target lesion is in an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
* The lesion requires treatment other than percutaneous transluminal angioplasty (PTA) prior to stent placement;
* Other lesions requiring treatment or surgery within 30 days of the procedure (pre or post) with the exception of the non-target lesion(s).
* Inadequate distal run-off.
* History of bleeding diatheses or coagulopathy or will refuse blood transfusions;
* Creatinine > 2.5 mg/dl
* Platelet count <80,000 cells/mm3 or >700,000 cells/mm3, or a white blood cell (WBC) of <3,000 cells/mm3
* Participation in another investigational device or drug study and has not completed the primary endpoint(s) or that clinically interferes with the study endpoints;
* Previously enrolled in the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Molnar, MD, Principal Investigator — Michigan Vascular Research Center; William Gray, MD, Principal Investigator — NY Presbyterian Hospital
Locations (2):
- United States (2):
  - Michigan Vascular Research Center, Flint, Michigan
  - NY Presbyterian Hospital, New York, New York

REFERENCES:
- [Derived] Molnar RG, Gray WA; ACTIVE Trial Investigators. Sustained patency and clinical improvement following treatment of atherosclerotic iliac artery disease using the Assurant cobalt iliac balloon-expandable stent system. J Endovasc Ther. 2013 Feb;20(1):94-103. doi: 10.1583/12-4010.1. PMID 23391088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was for a period of 16 months. Subjects were recruited at medical clinics who participate in clinical trials.
Groups:
- Assurant Cobalt Iliac Stent: Cobalt stent implanted using standard percutaneous intervention technique.
Period: Overall Study
Arm/Group | Assurant Cobalt Iliac Stent
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Assurant Cobalt Iliac Stent: Treatment with iliac stenting
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 65.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 69
Region of Enrollment [Number; unit: participants]
  United States | 123

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events (MAE), Measured as Device and/or Procedure Related Death, Target Limb Loss and/or Clinically Driven Target Lesion Revascularization (TLR) or Target Vessel Revascularization (TVR).
Description: Percentage based on number of evaluable subjects for MAE. Subjects are considered unevaluable for MAE to 9 months if a) withdrawn before 240 days without having MAE events or b) lost to follow-up before 240 days without having MAE events and had no contact thereafter or c) any device and/or procedure-unrelated death before 240 days without having MAE events.
Time Frame: 9 months
Population: Intent to Treat population (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
percentage of participants | 0.8 [0 to 4.5]

2. Secondary Outcome: Primary Patency Rate at 9 Months
Description: Primary patency was defined as the blood flow through the treated vessel segment into the distal vasculature (e.g. the common femoral artery and/or the deep femoral artery) as evidenced by duplex ultrasound scan at 9 months for all subjects enrolled with evaluable duplex scans.
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Lesions) | 141
percentage of lesions | 100

3. Secondary Outcome: Device Success
Description: Device Success defined as angiographic evidence of <30% final residual stenosis of the target lesion using only the assigned device.
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesion
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Lesion) | 159
percentage of lesions | 97.5 [0 to 0]

4. Secondary Outcome: Lesion Success
Description: Lesion Success defined as angiographic evidence of <30% final residual stenosis of the target lesion using any percutaneous method such as baloon angioplasy or other stent.
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Lesions) | 159
percentage of lesions | 97.5

5. Secondary Outcome: Procedure Success
Description: Procedure Success defined as angiographic evidence of <30% final residual stenosis of the target lesion after stent placement and no occurrence of a procedure related MAE prior to hospital discharge (for subjects with more than one lesion stented the worse case is counted)
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of participants
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
percentage of participants | 96.7

6. Secondary Outcome: Clinical Success
Description: Clinical success defined as the improvement of Fontaine classification by at least one stage above the pretreated (pre-procedure) clinical value. The reported values are a percentage of limbs showing improvement.
Time Frame: 30 days
Population: Intent to Treat population
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Limbs) | 152
percentage of limbs | 88.2

7. Secondary Outcome: Clinical Success
Description: as for outcome 6
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Limbs) | 146
percentage of limbs | 90.4 [84.4 to 94.7]

8. Secondary Outcome: Hemodynamic Success
Description: Hemodynamic success defined as an improvement in ankle-brachial Index (ABI) or toe brachial index (TBI) > 0.10 over pre-procedure level and not deteriorated by > 0.15 from first post-procedure level.
Time Frame: 30 days
Population: Intent to Treat population
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Limbs) | 153
percentage of limbs | 64.1

9. Secondary Outcome: Hemodynamic Success
Description: as for outcome 8
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
Number analyzed (Limbs) | 143
percentage of limbs | 55.2

10. Secondary Outcome: All Cause Mortality
Description: Subjects are considered unevaluable for all cause mortality at 30 days if a) withdrawn before 25 days or b) lost to follow-up before 25 days and had no contact thereafter.
Time Frame: 30 days
Population: Intent to Treat population
Measure: Number; unit: participants
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 123
participants | 0.0

11. Secondary Outcome: All Cause Mortality
Description: Subjects are considered unevaluable for all cause mortality at 9 months if a) withdrawn before 240 days or b) lost to follow-up before 240 days and had no contact thereafter.
Time Frame: 9 months
Population: Intent to Treat population
Measure: Number; unit: participants
Arm/Group | Assurant Cobalt Iliac Stent
Number analyzed (Participants) | 121
participants | 0.0 [0 to 3.0]

ADVERSE EVENTS:
Time Frame: From subject index procedure through the 9 month follow up visit period.
Groups:
- Assurant Cobalt Iliac Stent: Treatment with Iliac stenting system
Arm/Group | Assurant Cobalt Iliac Stent
Serious Adverse Events (participants affected / at risk) | 37/123
Other Adverse Events (participants affected / at risk) | 78/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assurant Cobalt Iliac Stent (N=123)
GASTROINTESTINAL DISORDERS (Vascular disorders) | 2 (2)
CARDIAC DISORDERS (Cardiac disorders) | 14 (14)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 3 (3) — General disorders and administration site conditions are not stent site disorders/complicatons rather site access point condition due to sheath introduction.
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 8 (8)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 5 (5)
INVESTIGATIONS (Investigations) | 1 (1)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS (Musculoskeletal and connective tissue disorders) | 5 (5)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 3 (3)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
VASCULAR DISORDERS (Vascular disorders) | 15 (15)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assurant Cobalt Iliac Stent (N=123)
CARDIAC DISORDERS (Vascular disorders) | 20 (20)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 14 (14)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 17 (17)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 17 (17)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 14 (14)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 8 (8)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS (Musculoskeletal and connective tissue disorders) | 22 (22)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 8 (8)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 9 (9)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 11 (11)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 9 (9)
VASCULAR DISORDERS (Vascular disorders) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medtronic has a legitimate interest in ensuring that a multi-center publication is the first publication to be released regarding the completed Study. The Institution agrees that it will not publish or disclose any results of or information pertaining to the study until a multi-center publication is released. If a publication is not released within one year after completion of the study, the Institution will have the right to publish information pertaining to their activities conducted.